CLINICAL TRIAL: NCT06389253
Title: Subtalar Extra-articular Screw Arthroereisis: How Does the Screw Work
Brief Title: Subtalar Extra-articular Screw Arthroereisis
Status: Not yet recruiting | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Professor Giacomo Placella, Professor, Università Vita-Salute San Raffaele
Other Study IDs: HTSW1
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Flatfoot, Flexible
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Control group are patients that will insert the calcaneo-stop screw (age between 10 and 14 years old).
  Interventions: Other: Histological Analysis
- Study Group: Study group are patient that remove the calcaneo-stop screw (age from 14 years old)
  Interventions: Other: Histological Analysis

INTERVENTIONS:
Other: Histological Analysis — For the study, a minimal part of the periarticular tissue, specifically the sinus tarsi juxta-articular fatty tissue, that is normally dissected and discarded during the surgical operation of insertion and removal of the calcaneo-stop screw, will be analyzed

SUMMARY:
The aim of the study is to investigate the effect of subtalar extra-articular calcaneo-stop screw on the proprioceptive and nociceptive pathways of the ankle before and after implantation. The hypothesis of the study is that an increased number of receptors related to proprioception will be detected in the sinus tarsi.

ELIGIBILITY:
Inclusion Criteria:

Study Group:

* Patients aged 14 years old and above that will remove the calcaneo stop screw, in place for at least 3 years after the implant, will be recruited
* Patients willing and able to give informed consent for the participation in the study. For underage patients, a parent/legal representative will give consent for the participation in the study.
* Male and female patients in fertile age can be recruited.

Control Group:

* Syndromic patients
* Previous foot malformation (synostosis, congenital clubfoot)
* Female participant who is pregnant, lactating or planning pregnancy during the course of the study.

Exclusion Criteria:

Control Group:

* Syndromic patients
* Previous foot malformation (synostosis, congenital clubfoot)
* Female participant who is pregnant, lactating or planning pregnancy during the course of the study.

Study Group:

* Patients suffering from post-operative complications
* Syndromic patients
* Previous foot malformation (synostosis, congenital clubfoot)
* Female participant who is pregnant, lactating or planning pregnancy during the course of the study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with subtalar extraarticular screw arthroereisis, gender male and female, no comorbidities.
  Control group are patients that will insert the calcaneo-stop screw (age between 10 and 14 years old).
  Study group are patient that remove the calcaneo-stop screw (age from 14 years old)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint (%) | Time 0 (baseline)
  Percentage of patients presenting at least one proprioceptive fibers in the pericapsular tissue

SECONDARY OUTCOMES:
Secondary Endpoint | Time 0 (baseline)
  Number and type of nervous fibers

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ircss Ospedale San Raffaele, Milan, Lombardy
  - Università Vita-Salute San Raffaele, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Pellegrin M, Moharamzadeh D. Subtalar Arthroereisis for Surgical Treatment of Flexible Flatfoot. Foot Ankle Clin. 2021 Dec;26(4):765-805. doi: 10.1016/j.fcl.2021.07.007. Epub 2021 Oct 4. PMID 34752238
- [Background] Michaudet C, Edenfield KM, Nicolette GW, Carek PJ. Foot and Ankle Conditions: Pes Planus. FP Essent. 2018 Feb;465:18-23. PMID 29381041
- [Background] Mosca VS. Flexible flatfoot in children and adolescents. J Child Orthop. 2010 Apr;4(2):107-21. doi: 10.1007/s11832-010-0239-9. Epub 2010 Feb 18. PMID 21455468
- [Background] Harris EJ. The natural history and pathophysiology of flexible flatfoot. Clin Podiatr Med Surg. 2010 Jan;27(1):1-23. doi: 10.1016/j.cpm.2009.09.002. PMID 19963167
- [Background] Jane MacKenzie A, Rome K, Evans AM. The efficacy of nonsurgical interventions for pediatric flexible flat foot: a critical review. J Pediatr Orthop. 2012 Dec;32(8):830-4. doi: 10.1097/BPO.0b013e3182648c95. PMID 23147627
- [Background] De Pellegrin M, Moharamzadeh D, Strobl WM, Biedermann R, Tschauner C, Wirth T. Subtalar extra-articular screw arthroereisis (SESA) for the treatment of flexible flatfoot in children. J Child Orthop. 2014 Dec;8(6):479-87. doi: 10.1007/s11832-014-0619-7. Epub 2014 Nov 21. PMID 25413354
- [Background] Rein S, Manthey S, Zwipp H, Witt A. Distribution of sensory nerve endings around the human sinus tarsi: a cadaver study. J Anat. 2014 Apr;224(4):499-508. doi: 10.1111/joa.12157. Epub 2014 Jan 29. PMID 24472004
- [Background] Freeman MA, Wyke B. The innervation of the knee joint. An anatomical and histological study in the cat. J Anat. 1967 Jun;101(Pt 3):505-32. No abstract available. PMID 6051731
- [Background] Hagert E, Forsgren S, Ljung BO. Differences in the presence of mechanoreceptors and nerve structures between wrist ligaments may imply differential roles in wrist stabilization. J Orthop Res. 2005 Jul;23(4):757-63. doi: 10.1016/j.orthres.2005.01.011. Epub 2005 Mar 29. PMID 16022987
- [Background] Hagert E. Proprioception of the wrist joint: a review of current concepts and possible implications on the rehabilitation of the wrist. J Hand Ther. 2010 Jan-Mar;23(1):2-17. doi: 10.1016/j.jht.2009.09.008. Epub 2009 Dec 5. PMID 19963343